CLINICAL TRIAL: NCT06319937
Title: The Role of Muscle Architecture as a Determinant of Functional Performance in Women With Knee Osteoarthritis
Brief Title: Muscle Architecture in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, PT, PhD, Prof., Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OA2023
Record Dates: First submitted 2024-01-26; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis; Foot Deformities; Muscle Weakness; Kinesiophobia
Keywords: knee osteoarthritis; ultrasonography; kinesiophobia; functional performance; muscles; foot
MeSH Terms: conditions — Osteoarthritis, Knee; Foot Deformities; Muscle Weakness; Kinesiophobia | interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OA Group (Experimental): Knee OA were included in the study. All patients exhibited evident radiographic changes in either unilateral or bilateral knees, consistent with a diagnosis of osteoarthritis, and were classified as Kellgren Lawrence (K-L) grade 2.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound

SUMMARY:
Background: The aim of this study was to compare the knee and ankle muscle architecture and plantar pressure distribution differences in knee osteoarthritis (OA) women with healthy women.

Methods: Fifty women with knee OA (Mean age=52.11±4.96 years, mean BMI=30.94±4.23 kg/m2) and fifty healthy women (Mean age= 50.93±3.78 years, mean BMI=29.06±4.82 kg/m2) were included in the study. Ultrasonography was used to evaluate Rectus Femoris (RF), Vastus Medialis (VM), Vastus Lateralis (VL), Peroneus Longus (PL), Tibialis Anterior (TA), and Medial Gastrocnemius (MG) muscle thickness, pennation angle, fascicle length, and fat thickness. The plantar pressure distribution was evaluated using the Digital Biometry Scanning System and software (DIASU, Italy).

DETAILED DESCRIPTION:
The following measurements were performed in subjects with knee osteoarthritis and healthy subjects with similar age-BMI and then a comparison was made between the 2 groups.

Measurements Pain severity: The Visual Analogue Scale (VAS) was used to assess the severity of knee and foot pain during activity. The 10-cm horizontal line was defined as 0 "no pain" and 10 "very severe pain", and the patients were asked to indicate their knee and foot pain level by drawing a line. This line was then measured in centimeters on both the dominant and non-dominant side.

Static foot posture: The Foot Posture Index (FPI) was used to evaluate foot posture in a relaxed position while standing. The FPI is showed to be a valid and reliable tool in individuals with knee OA. The FPI consisted of six items: 1) palpation of the talar head, 2) assessment of the curvature of the supra and infra lateral malleolus, 3) evaluation of the frontal plane position of the calcaneus, 4) identification of any prominence in the region of the talonavicular joint, 5) examination of the congruence of the medial longitudinal arch, and 6) measurement of abduction/adduction of the forefoot on the rear foot. Each item was scored from -2 to +2, and the total score ranged from -12 to +12. A higher positive score indicated a more pronated foot. A score of ≥6 indicated a pronated foot type, while scores of 0-5 indicated a neutral foot type, and scores of ≤-1 indicated a supinated foot type. OA side and dominant side assessed. All data on static foot posture were collected by the physiotherapist who has 5 years of experience in foot assessment (X). To avoid bias, the physiotherapist performing the assessment did not know which group the individuals were in.

Muscle architecture: Ultrasound, which is a measurement method with validity and reliability in individuals with knee OA, was used to evaluate the knee and ankle muscles. A total of six muscles were evaluated, including three knee muscles and three ankle muscles: Rectus Femoris (RF), Vastus Medialis (VM), Vastus Lateralis (VL), Tibialis Anterior (TA), Peroneus Longus (PL) and Medial Gastrocnemius (MG). The muscle thickness, pennation angle, fascicle length and fat thickness of each muscle were evaluated using B-Mode ultrasonography (E-Saote MyLab X8 eXP Ultrasound System, Florence, Italy) and a linear array transducer (4-11.4 MHz). It has been mentioned that there is muscle weakness in the muscles around the knee in knee OA, and in line with the investigators' hypothesis, the investigators thought that there may be differences in the muscles around the foot in these patients, so the investigators preferred to evaluate these muscles. All data on muscle architecture were collected by the same rheumatologist who has 5 years of experience in ultrasound assessment.

The images of the RF, VM, VL, and TA muscles were obtained with participants in a supine position. For the MG and PL muscle images, participants were instructed to lie prone. To enhance reproducibility and minimize the risk of sampling a muscle obliquely, the transducer was oriented parallel to the muscle fascicles and perpendicular to the skin.

The image was regarded as optimized when a thin layer of gel was visible between the skin and the transducer, signifying that no manual compressive forces were distorting the muscle after it had been identified. The same researcher then slightly retracted the transducer to avoid compressing the muscle. Ultrasound images were analyzed using Image J program (Version 1.53p, 2022, National Institutes of Health, Bethesda, MD, USA) by the same researcher. The same procedure was employed for each muscle group, with measurements taken of both muscle architecture and fat thickness. Following completion of all images from the first extremity, the identical technique was utilized to image the opposite lower extremity. Muscle thickness was measured as the distance between the internal borders of the superficial and deep aponeuroses. Fat thickness of all muscles was measured as the distance between the skin of the superficial aponeuroses. Pennation angle was defined as the angle between the muscle fascicle line and the deep aponeuroses. Fascicle length was defined as the distance between the origin of the fascicle at the superficial aponeuroses and insertion of the same fascicle in the deep aponeuroses.

Femoral cartilage thickness: In order to determine femoral cartilage thickness, individuals assumed a supine position with their knees comfortably flexed to the maximum extent. The probe was positioned axially on the suprapatellar region. Femoral cartilage thickness was assessed at three discrete points on both knees, specifically at the levels of the lateral condyle, intercondylar area, and medial condyle. Water-soluble gel was applied between the transducer and the skin to support acoustic coupling, without applying pressure to the muscle. The transducer was oriented axially above the patellar outer edge. In addition, femoral cartilage thickness measurement is a valid and reliable measurement.

Plantar pressure distribution: Plantar pressure distribution was performed by the Digital Biometric Images Scanning System and relevant Milletrix software (Diagnostic Support; Diasu Health Technologies, Rome, Italy). The platform employed in this study comprised a 5-meter long and 40-centimeter wide walkway equipped with 4024 sensors that could sample data at a frequency of 300 MHz. The force platform assessed plantar pressure on both feet while standing, and it calculated the average percentage of pressure distribution for each foot. Participants were instructed to stand barefoot on the platform for 10 seconds, facing a reference point, with their arms hanging comfortably by their sides. During these measurements, the patients were instructed not to consciously adjust their posture.

The static evaluation provided information on numerical surface and loading values, both globally (for each foot) and partially (relative to the rearfoot, forefoot, medial and lateral load). The maximum foot pressure (FPmax), average foot pressure (Pavg.), total surface area, forefoot load (FFL), rearfoot load (RFL), total load on the foot, medial load, lateral load, foot angle (FA) and foot progression angle (FPA) of the women were recorded. Foot angle is the angle between the direction of progression of the individual and a reference line on the sole of each foot. Foot progression angle is the angle between the longitudinal foot axis and the vertical axis of the foot. The plantar pressure distribution outcomes of the related knee in patients with unilateral involvement and the most symptomatic knee in patients with bilateral knee involvement were compared with matched knees of the healthy controls . To ensure blinding in the study, plantar pressure distribution was performed by a physiotherapist with 7 years of experience in this field. To avoid bias, the physiotherapist performing the assessment did not know which group the individuals were in.

Kinesiophobia: The Tampa Kinesiophobia Scale (TKS) was used to assess fear of movement-related pain. This scale, consisting of twenty-three items, assesses the inhibition or fear of movement due to feelings of vulnerability caused by painful conditions. The total score ranges from 17 to 68 points. A high score on the scale indicates a high level of kinesiophobia.

Functional Performance : Functional performance was assessed using the stair-climbing test (SCT) and the 10-time sit-stand test (SST), which were approved for use in individuals with KOA and recommended by the International Osteoarthritis Research Association. For the SCT, individuals were asked to ascend, turn around, and descend a flight of 10 steps as quickly as possible, using one handrail if necessary. The time to ascend and descend was measured. For the SST, individuals were asked to stand up completely straight from a chair with armrests, and sit down again without support from their arms, and repeat this 10 times at the fastest pace they could. The time during this procedure was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-65 years
* Activity-related knee pain
* Morning knee stiffness for 30 min
* Knee pain on most days for 3 months or more

Exclusion Criteria:

* Having lower extremity surgery
* Conditions that cause congenital or developmental diseases
* The presence of systemic inflammatory arthritis
* Polyneuropathy/lower extremity neuropathy, severe radiculopathy
* Having undergone physical therapy, exercises or knee injections for the knee in the previous 6 months
* Congenital foot deformity
* BMI higher than 35 kg/m2

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | 15 days
  Muscle thickness of Rectus Femoris, Vastus Medialis, Vastus Lateralis, Medial Gastrocnemius, Peronalis Longus.
  Muscle thickness of Rectus Femoris, Vastus Medialis, Vastus Lateralis, Medial Gastrocnemius, Peronalis Longus.
  Ultrasound, which is a measurement method with validity and reliability in individuals with knee OA, was used to evaluate the knee and ankle muscles. A total of six muscles were evaluated, including three knee muscles and three ankle muscles: Rectus Femoris (RF), Vastus Medialis (VM), Vastus Lateralis (VL), Tibialis Anterior (TA), Peroneus Longus (PL) and Medial Gastrocnemius (MG). The muscle thickness of each muscle were evaluated using B-Mode ultrasonography (Esaote MyLab X8 eXP Ultrasound System, Florence, Italy) and a linear array transducer (4-11.4 MHz)
Pennation angle | 15 days
  Pennation angle of Rectus Femoris, Vastus Medialis, Vastus Lateralis, Medial Gastrocnemius, Peronalis Longus.
  Ultrasound, which is a measurement method with validity and reliability in individuals with knee OA, was used to evaluate the knee and ankle muscles. A total of six muscles were evaluated, including three knee muscles and three ankle muscles: Rectus Femoris (RF), Vastus Medialis (VM), Vastus Lateralis (VL), Tibialis Anterior (TA), Peroneus Longus (PL) and Medial Gastrocnemius (MG). The pennation angle of each muscle were evaluated using B-Mode ultrasonography (Esaote MyLab X8 eXP Ultrasound System, Florence, Italy) and a linear array transducer (4-11.4 MHz)
Fat thickness | 15 days
  Fat thickness of Rectus Femoris, Vastus Medialis, Vastus Lateralis, Medial Gastrocnemius, Peronalis Longus.
  Ultrasound, which is a measurement method with validity and reliability in individuals with knee OA, was used to evaluate the knee and ankle muscles. A total of six muscles were evaluated, including three knee muscles and three ankle muscles: Rectus Femoris (RF), Vastus Medialis (VM), Vastus Lateralis (VL), Tibialis Anterior (TA), Peroneus Longus (PL) and Medial Gastrocnemius (MG). The fat thickness of each muscle were evaluated using B-Mode ultrasonography (Esaote MyLab X8 eXP Ultrasound System, Florence, Italy) and a linear array transducer (4-11.4 MHz)

SECONDARY OUTCOMES:
Stair climbing test | 15 days
  Functional performance was assessed using the stair-climbing test (SCT) time which were approved for use in individuals with KOA and recommended by the International Osteoarthritis Research Association. For the SCT, individuals were asked to ascend, turn around, and descend a flight of 10 steps as quickly as possible, using one handrail if necessary. The time to ascend and descend was measured.
Sit-stand test | 15 days
  Functional performance was assessed using the 10-time sit-stand test (SST), which were approved for use in individuals with KOA and recommended by the International Osteoarthritis Research Association. For the SST, individuals were asked to stand up completely straight from a chair with armrests, and sit down again without support from their arms, and repeat this 10 times at the fastest pace they could. The time during this procedure was recorded.